CLINICAL TRIAL: NCT07352969
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, 24 Months Treatment Duration, Dose Finding Study, to Evaluate Efficacy, Safety and Pharmacodynamics of IBI3016 in Mild to Moderate Hypertensive Patients
Brief Title: A Dose Finding Study of IBI3016 in Mild to Moderate Hypertensive Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI3016A201
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- IBI3016 dose 4 (Experimental): subcutaneous injection
  Interventions: Drug: IBI3016
- IBI3016 dose 1 (Experimental): subcutaneous injection
  Interventions: Drug: IBI3016
- IBI3016 dose 2 (Experimental): subcutaneous injection
  Interventions: Drug: IBI3016
- placebo (Placebo Comparator): subcutaneous injection
  Interventions: Other: Placebo
- IBI3016 dose 3 (Experimental): subcutaneous injection
  Interventions: Drug: IBI3016
- IBI3016 dose 5 (Experimental): subcutaneous injection
  Interventions: Drug: IBI3016

INTERVENTIONS:
Drug: IBI3016 — Solution of Injection
  Arms: IBI3016 dose 1; IBI3016 dose 2; IBI3016 dose 3; IBI3016 dose 4; IBI3016 dose 5
Other: Placebo — 0.9% sodium chloride saline solution
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of IBI3016 or placebo, given subcutaneously, every 3 or 6 months, at different dose levels in patients with mild to moderate hypertension

DETAILED DESCRIPTION:
Phase 2, multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy, safety, and pharmacodynamics of IBI3016 in patients with mild to moderate hypertension. Multiple doses of IBI3016 will be tested against placebo, administered as subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Males or females aged 18 to 75 years.
3. Diagnosis of primary hypertension without anti-HTN medication or with one anti-HTN medication
4. Mean sitting SBP ≥140 mmHg and < 170 mmHg measured by OBPM.
5. Participants able to understand and comply with study procedures.

Exclusion Criteria:

1. Known history of secondary hypertension.
2. Orthostatic hypotension.
3. Laboratory parameter assessments outside of range at screening：

   * Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 2× Upper Limit of Normal (ULN)
   * Total Bilirubin > 1.5× ULN
   * International Normalized Ratio (INR) > 2.0
   * Serum Potassium > 5 mg/L
   * Estimated Glomerular Filtration Rate (eGFR) ≤ 45 mL/min/1.73m²
   * QTcF > 480 ms
4. Medical condition, other than hypertension, requiring treatment with RAAS inhibitor.
5. Current or history of intolerance to ACEi and/or ARBs.
6. Acute myocardial infarction (AMI), unstable angina, percutaneous coronary intervention (PCI) , coronary artery bypass graft (CABG), ischemic or hemorrhagic stroke, transient ischemic attack, or clinically significant cardiac arrhythmias within 6 months prior to screening. Any history of congestive heart failure.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2029-03-27 (Estimated); Study Completion 2029-03-27 (Estimated)

PRIMARY OUTCOMES:
Change in SBP by OBPM | From baseline through month 3
  Change from baseline at Month 3 in systolic blood pressure (SBP) by office blood pressure measurement (OBPM)

SECONDARY OUTCOMES:
Change in Mean 24hr SBP by ABPM | From baseline through month 3
  Change from baseline at Month 3 in mean 24hr SBP by ambulatory blood pressure measurement (ABPM)
Change in SBP and DBP by OBPM | From baseline through month 6
  Change from baseline through month 6 in SBP and diastolic blood pressure (DBP) by OBPM
Change in Mean 24hr, mean daytime, mean nighttime SBP and DBP by ABPM | Change from baseline through month 6 in Mean 24hr, mean daytime, mean nighttime SBP and DBP by OBPM
  From baseline through month 6
Percentage Change in AGT by blood test | From baseline through month 24
  Percentage Change from baseline through month 24 in Angiotensinogen (AGT) by blood test

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China